CLINICAL TRIAL: NCT02948205
Title: Analysis of Trans-umbilical Laparoendoscopic Single-site Surgery by 3D Laparoscopy in the Treatment of Infertility
Brief Title: Analysis of TU-LESS by 3D Laparoscopy in the Treatment of Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-3D
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Infertility, Female
Keywords: Infertility, TU-LESS, 3D laparoscopy
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3D group (Experimental): infertility patient get TU-LESS by 3D Laparoscopy
  Interventions: Procedure: 3D group
- normal group (Other): infertility patient get normal laparoscopic surgery
  Interventions: Procedure: normal group

INTERVENTIONS:
Procedure: 3D group — infertility patient get TU-LESS by 3D Laparoscopy
  Arms: 3D group
Procedure: normal group — infertility patient get normal laparoscopic surgery
  Arms: normal group

SUMMARY:
This study intends to carry out a prospective, randomized controlled trial to compare the trans-umbilical laparoendoscopic single-site surgery by 3D laparoscopy with normal laparoendoscopic surgery in the treatment of infertility patient, so as to further clarify the safety and curative effect of TU-LESS by 3D laparoscopy and provide evidence-based basis for its application in infertility population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are younger than 36 and older than 24.
2. Clearly diagnosed with female Infertility.
3. Infertility within 1 to 10 years.
4. informed consent form signed

Exclusion Criteria:

1. Over the age of 35.
2. Indefinite diagnosis.
3. With severe medical problems (severe liver disease, kidney disease, respiratory diseases, heart disease or uncontrolled diabetes, epilepsy, etc., dysfunction of important organs).
4. abdominal surgery history
5. Unwilling to comply with the research plan.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
pain score | in 24 hours after surgery
  Visual Analogue Score for the pain feeling of the patient
pregnancy rate | 6 months after surgery

SECONDARY OUTCOMES:
Operation time | intraoperative

IPD SHARING:
Plan to Share IPD: No